CLINICAL TRIAL: NCT07131124
Title: Can Selfcompassion Training Reduce Alcohol Consumption in Patients With Alcohol Use Disosrder ? Randomized Controlled Trial
Brief Title: Can Selfcompassion Training Reduce Alcohol Consumption in Patients With Alcohol Use Disosrder ?
Acronym: COMPAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Etablissement Public de Santé Barthélemy Durand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23P04; 2025-A00584-45 (Other: ANSM)
Record Dates: First submitted 2025-08-07; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Addiction; Addiction Disorders; Alcohol Use Disorders; Alcohol Dependence
Keywords: Self-compassion; Alcohol Use Disorders
MeSH Terms: conditions — Behavior, Addictive; Alcoholism | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Self-Compassion (MSC) program + Treatment As Usual (TAU) (Experimental): Participants in this group will attend 9 group sessions of the Mindful Self-Compassion (MSC) program in addition to 9 sessions of Treatment As Usual (TAU), for a total of 18 sessions during the intervention period.
  Interventions: Behavioral: Mindful Self-Compassion program; Behavioral: Treatment As Usual (TAU) program
- Treatment As Usual (TAU) (Active Comparator): Participants in this group will attend 18 sessions of Treatment As Usual (TAU) during the intervention period.
  Interventions: Behavioral: Treatment As Usual (TAU) program

INTERVENTIONS:
Behavioral: Mindful Self-Compassion program — The MSC self-compassion program will be delivered by instructors trained by the LBCM Organization, certified Qualiopi and affiliated to the ADM (accredited training organization).
  The MSC program consists of 8 weekly sessions, each 2.5 hours long, plus an additional half-day of supplementary practice .
  Arms: Mindful Self-Compassion (MSC) program + Treatment As Usual (TAU)
Behavioral: Treatment As Usual (TAU) program — Current treatment strategies for Alcohol Use Disorders (AUD) rely on a combination of pharmacological and psychotherapeutic treatments (Schuckit, 2009). The three specialized outpatient centers participating in our study provide comprehensive and up-to-date addiction care that meets international and national recommendations (HAS, 2023; SFA, 2023).
  The services offered, in addition to standard care, include:
  Brief interventions, Psychoeducation sessions, Motivational interview, Individual and group therapies for patients (cognitive-behavioral therapies, cognitive remediation, relaxation techniques), Individual and group therapies for families, Psychosocial interventions, including social support and strengthening of psychosocial skills, Peer support groups (peer helpers, expert patients, former user groups)

SUMMARY:
The objective of this interventional study is to evaluate the effectiveness of the Mindful Self-Compassion (MSC) program in reducing alcohol consumption in a population of individuals with Alcohol Use Disorder (AUD), six months after the intervention. The MSC program was designed to enhance self-compassion skills. It has demonstrated a mediating effect on symptoms of stress, depression, and anxiety, which are known to contribute to the maintenance of AUD.

Outpatients with AUD will be included after providing informed consent and will be randomized into two groups (MSC+TAU vs TAU). The follow-up includes 13 visits over a 9-month period, with group sessions according to allocation. Three follow-up visits are scheduled up to six months after the end of the sessions. Participants will complete several scales and surveys (AUDIT, TLFB, SCS, HAD, SSS-S, TOSCA-3, AQoLS, MAAS, Fagerström, CUDIT-R, EVA craving).

DETAILED DESCRIPTION:
Context:

Alcohol Use Disorders (AUD, ICD-10, DSM-5) affect more than 11% of men and 3% of women in France, leading to over 200 diseases and 41,000 deaths annually, primarily due to alcohol-related cancers. The current management of patients with AUD is based on a combination of pharmacological and psychotherapeutic treatments. However, 60% of patients at 6 months and 70% at 1 year fail to significantly reduce their alcohol consumption or maintain abstinence. Therefore, it is crucial to explore new complementary therapeutic strategies.

Self-compassion involves treating oneself with the same kindness, attention, and understanding that we extend to others in times of suffering. Several studies suggest that self-compassion is a key factor in promoting proactive health behaviors and improving adherence in conditions such as diabetes, HIV-related illnesses, and schizophrenia. Individuals with AUD tend to have lower levels of self-compassion compared to the general population, whereas higher levels of self-compassion have shown protective effects against the development and persistence of AUD.

Objectives :

The primary objective is to evaluate the effectiveness of the Mindful Self-Compassion (MSC) program in reducing alcohol consumption among individuals with AUD, measured by the number of heavy drinking days assessed using the Timeline Follow-Back (TLFB) method, six months after treatment completion.

The secondary objectives include evaluating the impact of the MSC program on reducing alcohol consumption by comparing the number of heavy drinking days at one and three months, as well as the total number of drinking days at one, three, and six months between groups using the TLFB method. Biomarkers CDT and GGT will be analyzed at one, three, and six months post-intervention to compare blood values.

The program's impact on psychological and behavioral factors will also be assessed using standardized scales at one, three, and six months.

Finally, program satisfaction and adherence will be measured using the CSQ-8 scale, session attendance rates, and the percentage of program completion (≥6/8 MSC sessions).

Research Hypothesis :

Alcohol consumption will be significantly reduced in the group of patients who complete the MSC program compared to the group receiving only standard treatment (Treatment As Usual: TAU).

Method :

This is a prospective, randomized, controlled, multicenter, single-blind, parallel-group interventional study RIPH2 (French interventional research category). The study follows the CONsolidated Standards of Reporting Trials (CONSORT) 2010 guidelines, updated in 2025.

Adult outpatients with AUD (ICD-10 and DSM-5 criteria) will be included after verification of eligibility criteria and the collection of informed consent. Participants will be randomized to one of the following groups:

* MSC+TAU group: receiving self-compassion training with the MSC program in addition to standard treatment
* TAU group: receiving only standard treatment Each participant will complete 13 visits over 9 months. The MSC+TAU group will attend 9 MSC sessions and 9 TAU sessions (18 sessions in total), while the TAU group will attend 18 TAU sessions. Follow-up assessments will take place at 1, 3, and 6 months after the final session. Participants will exit the study after 245 days (9 months) of follow-up.

The study aims to recruit 152 participants over 24 months across three centers (EPS Barthélemy Durand, Paul Brousse University Hospital, EPSM de l'Oise, CHI Montdidier), with an expected start date of October 2025 and a total study duration of 36 months.

Expected public health impact :

Self-compassion training with the MSC program is expected to significantly reduce alcohol consumption in individuals with AUD. If the results are positive, the MSC program could facilitate alcohol reduction, potentially lowering the risk of alcohol-related disorders, particularly alcohol-induced cancers (e.g., larynx, pharynx, esophagus, breast, liver, bladder, etc.).

Perspectives :

If effective, the MSC self-compassion training program could be implemented in clinical practice to help patients with AUD who are not yet ready to quit drinking but need a supportive approach to reduce their alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years.
* Subjects meeting DSM-5 criteria for Alcohol Use Disorder (AUD).
* Subjects receiving outpatient care in addiction services, CSAPA, CMP, day hospitals, mental health care institutions, community mental health centers.
* Subjects affiliated with the social security system.
* Subjects who have a good understanding of French languague, allowing them to provide informed consent, respond to self-questionnaires, and participate in the MSC program.

Exclusion Criteria:

* Subjects unable to understand the questionnaires.
* Subjects presenting moderate or severe suicidal ideation (assessed by the Suicide item of the MINI scale).
* Subjects with a score <10 on the MoCA version 7.1 test.
* Subjects admitted to inpatient units (since hospitalization alters alcohol consumption).
* Subjects unable to provide informed or voluntary consent to participate in the study.
* Subjects under guardianship or curatorship.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Assess the effectiveness of the Mindful Self-Compassion (MSC) program in reducing alcohol consumption in a population with Alcohol Use Disorder (AUD) six months after the intervention | 6 months
  The primary outcome measure is the number of heavy drinking days, assessed using the Timeline Follow-Back (TLFB) method, six months after the end of treatment, in both the MSC+Treatment as Usual (TAU) intervention group and the TAU control group

SECONDARY OUTCOMES:
Assess the effectiveness of the MSC program in reducing alcohol consumption in a population of individuals with AUD one and three months after the intervention. | 1 months, 3 months
  Comparison of the number of heavy drinking days, assessed using the TLFB method, one and three months after the intervention between the MSC+TAU and TAU groups.
Assess the effectiveness of the MSC program in reducing the number of alcohol consumption days in a population of individuals with AUD one, three, and six months after the intervention. | 1 months, 3 months, 6 months
  Comparison of the number of alcohol consumption days, assessed using the TLFB method, one, three, and six months after the intervention between the MSC+TAU and TAU groups.
Assess the effectiveness of the MSC program in reducing alcohol consumption in a population of individuals with AUD one, three, and six months after the intervention. | 1 months, 3 months, 6 months
  Comparison of blood levels of the biological markers Carbohydrate-Deficient Transferrin (CDT), one, three, and six months after the intervention between the MSC+TAU and TAU groups.
Assess the effectiveness of the MSC program in reducing alcohol consumption in a population of individuals with AUD one, three, and six months after the intervention. | 1 months, 3 months, 6 months]
  Comparison of blood levels of the biological marker Gamma-Glutamyl Transferase (GGT), one, three, and six months after the intervention between the MSC+TAU and TAU groups.
Evaluate the effectiveness of the MSC program on mean scores for the Alcohol Use Disorders Identification Test (AUDIT) in a population of individuals with AUD one, three, and six months after the intervention. | 1 month, 3 month, 6 month
  Comparison of mean scores obtained on the Alcohol Use Disorders Identification Test (AUDIT, French translation by Gache et al., 2005) at one, three, and six months after the intervention in the MSC+TAU and TAU groups.
Evaluate the effectiveness of the MSC program on self-compassion levels in a population of individuals with AUD, at one, three, and six months after the intervention. | 1 month, 3 month, 6 month
  Comparison of mean scores obtained on the Self-Compassion Scale (SCS, French translation by Kotsou et al., 2016) at one, three, and six months after the intervention between the MSC+TAU and TAU groups.
Evaluate the effectiveness of the MSC program on depression and anxiety levels in a population of individuals with AUD, at one, three, and six months after the intervention. | 1 month, 3 month, 6 month
  Comparison of mean scores obtained on the Hospital Anxiety and Depression Scale (HAD, French translation by Lepine et al., 2000) at one, three, and six months after the intervention between the MSC+TAU and TAU groups.
Evaluate the effectiveness of the MSC program on self-stigmatization levels in a population of individuals with AUD, at one, three, and six months after the intervention. | 1 month, 3 month, 6 month
  Comparison of mean scores obtained on the Self-Stigma Scale - Short Form (SSS-S, French translation by Golay et al., 2022) at one, three, and six months after the intervention between the MSC+TAU and TAU groups.
Evaluate the effectiveness of the MSC program on shame and guilt levels in a population of individuals with AUD, at one, three, and six months after the intervention. | 1 month, 3 month, 6 month
  Comparison of mean scores obtained on the Test of Self-Conscious Affect evaluating shame and guilt (French-TOSCA-3, French translation by Nugier et al., 2012) at one, three, and six months after the intervention between the MSC+TAU and TAU groups.
Evaluate the effectiveness of the MSC program on quality of life levels in a population of individuals with AUD, at one, three, and six months after the intervention. | 1 month, 3 month, 6 month
  Comparison of mean scores obtained on the Alcohol Quality of Life Scale (AQoLS, French translation by Luquiens et al., 2015) at one, three, and six months after the intervention between the MSC+TAU and TAU groups.
Evaluate the effectiveness of the MSC program on mindfulness levels in a population of individuals with AUD, at one, three, and six months after the intervention. | 1 month, 3 month, 6 month
  Comparison of mean scores obtained on the Mindfulness Attention Awareness Scale (MAAS, French translation by Jermann, 2009) at one, three, and six months after the intervention between the MSC+TAU and TAU groups.
Evaluate the effectiveness of the MSC program on craving levels in a population of individuals with AUD, at one, three, and six months after the intervention. | 1 month, 3 month, 6 month
  Comparison of mean scores obtained on the Visual Analog Scale for Craving (EVA, Mottola, 1993) at one, three, and six months after the intervention between the MSC+TAU and TAU groups.
Evaluate the effectiveness of the MSC program on tobacco use in a population of individuals with AUD, at one, three, and six months after the intervention. | 1 month, 3 month, 6 month
  Comparison of mean scores obtained on the Fagerström Test for Nicotine Dependence (Fagerström, French translation by WHO, Etter et al., 1999) at one, three, and six months after the intervention between the MSC+TAU and TAU groups.
Evaluate the effectiveness of the MSC program on cannabis use in a population of individuals with AUD, at one, three, and six months after the intervention. | 1 month, 3 month, 6 month
  Comparison of mean scores obtained on the Test of Cannabis Use Disorders Identification Test - Revised (CUDIT-R, French translation by Luquiens et al., 2021) at one, three, and six months after the intervention between the MSC+TAU and TAU groups.
Assess satisfaction with the MSC program among individuals with AUD. | 6 months
  Participant satisfaction, measured using the Client Satisfaction Questionnaire (CSQ-8)
Assess adherence to the MSC program among individuals with AUD. | 6 months
  Program adherence, assessed by the percentage of sessions attended by each participantn and Percentage of participants who completed the program, defined as attending at least 6 out of 8 sessions

CONTACTS AND LOCATIONS:
Overall Officials: Alain DERVAUX, Principal Investigator — Etablissement Public de Santé Barthélemy Durand
Locations (1):
- Etablissement Public de Santé Barthélemy Durand, Étampes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen, G. (2019). The Role of Self-Compassion in Recovery from Substance Use Disorders. Obm Icm, 4, 1-1.
- [Background] Fond G, Boyer L, Boucekine M, Aden LA, Schurhoff F, Tessier A, Andrianarisoa M, Berna F, Brunel L, Capdevielle D, Chereau I, Mallet J, Denizot H, Dorey JM, Dubertret C, Dubreucq J, Faget C, Gabayet F, Rey R, Richieri R, Passerieux C, Schandrin A, Urbach M, Vidailhet P, Llorca PM, Misdrahi D; FACE-SZ (FondaMental Academic Centers of Expertise for Schizophrenia) group. Validation study of the Medication Adherence Rating Scale. Results from the FACE-SZ national dataset. Schizophr Res. 2017 Apr;182:84-89. doi: 10.1016/j.schres.2016.10.023. Epub 2016 Oct 24. PMID 27789187
- [Background] Neff KD, Germer CK. A pilot study and randomized controlled trial of the mindful self-compassion program. J Clin Psychol. 2013 Jan;69(1):28-44. doi: 10.1002/jclp.21923. Epub 2012 Oct 15. PMID 23070875
- [Background] Neff KD. Self-Compassion: Theory, Method, Research, and Intervention. Annu Rev Psychol. 2023 Jan 18;74:193-218. doi: 10.1146/annurev-psych-032420-031047. Epub 2022 Aug 12. PMID 35961039